CLINICAL TRIAL: NCT03887923
Title: Vestibular Physical Therapy for People With Alzheimer Disease
Acronym: VPT in AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Brooke Klatt, Postdoctoral Fellow, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY18120038
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Vestibular Diseases; Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Vestibular Diseases; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular Physical Therapy (Experimental): Balance, Gaze Stabilization, Habituation, and Walking exercises
  Interventions: Behavioral: Vestibular Physical Therapy

INTERVENTIONS:
Behavioral: Vestibular Physical Therapy — Balance, Gaze Stabilization, Habituation, and Walking exercises
  Other Names: modified-Vestibular Physical Therapy

SUMMARY:
The purpose of this study is to assess the tolerability and preliminary efficacy of an 8-week home-based vestibular physical therapy program in people with cognitive impairment.

DETAILED DESCRIPTION:
This project uses a novel non-pharmacological treatment to improve balance and reduce falls in patients with Alzheimer Disease (AD) using a conceptual framework that combines current vestibular physical therapy (VPT) practice guidelines with the latest motor learning theories for cognitively-impaired patients. The modified VPT protocol for AD patients was developed by experts in VPT and motor learning in AD and will be tested. This pilot study will provide much-needed data about whether VPT can be adapted for patients with AD, and whether VPT shows promise in improving or stabilizing balance, spatial cognition, and gait function in patients with AD.

ELIGIBILITY:
Inclusion Criteria:

* mild-AD diagnosis
* complaints or observation of gat disturbance

Exclusion Criteria:

* inability to stand for 3 minutes without rest
* recent lower extremity fractures/severe sprains (within last six months)
* incapacitating back or lower extremity pain
* confounding neurologic or neuromuscular disorders
* presence of benign paroxysmal positional vertigo
* pain elicited during cervical range of motion or limited cervical range of motion

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Tolerability of Vestibular Physical Therapy in people with Alzheimer Disease: number of times modifications are needed to be made | 8 weeks
  The ability to perform the tasks within VPT will be monitored during each exercise within all eight training sessions. The number of times modifications are needed to be made to the protocol will be recorded (for example, the number of times the participant needs cuing to attend to the exercise for gaze stabilization which requires constant head movement for the 30-second exercise trial will be recorded).
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in balance performance for people with Alzheimer Disease; Gait velocity | 10 weeks (the outcomes will be obtained pre- and post-training)
  Gait velocity: preferred walking speed will be recorded over 10-meter distance and is measured in meters/second
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in balance performance for people with Alzheimer Disease: Four Square Step Test | 10 weeks (the outcomes will be obtained pre- and post-training)
  Four Square Step Test: dynamic balance, spatial, & sequencing skills will be assessed as participants step forward, backward, and sideways over a low obstacle and is measured by time (seconds) to complete the test
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in balance performance for people with Alzheimer Disease: Mini Balance Evaluation Systems Test | 10 weeks (the outcomes will be obtained pre- and post-training)
  Mini Balance Evaluation Systems Test: assesses anticipatory postural adjustment, reactive postural control, sensory orientation, and dynamic gait with a total score of 28

SECONDARY OUTCOMES:
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Montreal Cognitive Assessment | 10 weeks (the outcomes will be obtained pre- and post-training)
  Montreal Cognitive Assessment: assesses several cognitive domains and serves as a screening tool for detecting cognitive impairment with scores ranging from 0-30 (score over 26 is considered normal)
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Money Road Map Test | 10 weeks (the outcomes will be obtained pre- and post-training)
  Money Road Map Test assesses egocentric mental rotation in space by recording the total number of errors for right-left discrimination of mental rotation tasks.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Trail Making Test A | 10 weeks (the outcomes will be obtained pre- and post-training)
  Trail Making Test A: assesses executive function by recording the time to accurately connect a sequence of 25 consecutive targets on a sheet of paper.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Trail Making Test B | 10 weeks (the outcomes will be obtained pre- and post-training)
  Trail Making Test B: assesses visual attention and task switching by recording the time to accurately connect a sequence of 25 consecutive targets alternating between numbers and letters on a sheet of paper.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Digit Span Forward & Backward | 10 weeks (the outcomes will be obtained pre- and post-training)
  Digit Span Forward & Backward: assesses memory by recording how many digits the participant can repeat back in the correct order immediately after presentation
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Letter Fluency | 10 weeks (the outcomes will be obtained pre- and post-training)
  Letter Fluency: assesses verbal fluency by recording how many words that the participant can produce that begin with a certain letter in a 60-second timeframe.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Category Fluency | 10 weeks (the outcomes will be obtained pre- and post-training)
  Category Fluency: assesses verbal fluency by recording how many words that the participant can produce that are within a certain category in a 60-second timeframe.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Digit Symbol Substitution | 10 weeks (the outcomes will be obtained pre- and post-training)
  Digit Symbol Substitution assesses cognitive functioning by seeing how many correct digit-symbol pairs the participant can record in 90 seconds using a nine pair options.
Preliminary efficacy of an 8-week home-based Vestibular Physical Therapy program on change in cognitive function for people with Alzheimer Disease: Benton Visual Retention Test | 10 weeks (the outcomes will be obtained pre- and post-training)
  Benton Visual Retention Test: assesses visual perception and visual memory by asking participants to reproduce 10 different individual designs after a 10-second exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke N Klatt, PhD, PT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Alzheimer Disease Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No